CLINICAL TRIAL: NCT06128044
Title: A Phase 1, Multicenter, Open-Label Study of CB-012, a CRISPR-Edited Allogeneic Anti-CLL-1 CAR-T Cell Therapy in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CRISPR-Edited Allogeneic Anti-CLL-1 CAR-T Cell Therapy in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Acronym: AMpLify
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision - Pipeline Reprioritization
Sponsor: Caribou Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CB12A
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of CB-012 (Experimental): Part A (Dose Escalation) of CB-012 with increasing doses using a 3+3 design, during which the MTD and/or RDE will be identified.
  Interventions: Drug: CB-012
- Dose Expansion of CB-012 (Experimental): Part B (Dose Expansion) - participants will be enrolled to receive CB-012 at the RDE and/or MTD determined in Part A in order to the determine the RP2D.
  Interventions: Drug: CB-012

INTERVENTIONS:
Drug: CB-012 — CB-012 allogeneic CAR-T cell therapy targeting CLL-1 Cyclophosphamide and Fludarabine chemotherapy for lymphodepletion
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
CB-012 is an allogeneic chimeric antigen receptor (CAR-T) cell therapy that targets C-type lectin-like molecule-1 (CLL-1). This is a Phase 1 study to evaluate the safety, preliminary efficacy, and pharmacokinetics, of CB-012 (the study treatment) in adults with acute myeloid leukemia (AML) that has come back after prior treatment (relapsed) or did not respond or is no longer responding to other treatment (refractory). Participants must have received at least 1 but not more than 3 prior lines of treatment for AML .

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of AML with either refractory or relapsed disease,
* Non-proliferative disease
* No more than 3 prior lines of therapy (induction, consolidation with or without allogeneic stem cell transplant, and maintenance are considered 1 line of therapy)
* No available therapy with reasonable survival benefit
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 and fit for allogeneic stem cell transplant
* Adequate renal, hepatic, pulmonary, and cardiac function, with specific laboratory criteria
* Women of child-bearing potential and men with a female partner who has child-bearing potential must agree to use acceptable, effective methods of birth control.

Exclusion Criteria:

* Acute promyelocytic leukemia
* Extra-medullary disease (EMD) that is metabolically inactive by 18-FDG PET-CT
* Prior treatment with CAR-T cell therapy
* Allogeneic stem cell transplant within 100 days before lymphodepletion
* Active graft-vs-host disease requiring therapy
* Known active or prior history of central nervous system involvement
* Seropositive for or history of human immunodeficiency virus (HIV)
* Vaccinated with live, attenuated vaccine within 4 weeks prior to lymphodepletion
* Active hepatitis B or C infection
* Primary immunodeficiency or autoimmune disease
* Known life-threatening allergies, hypersensitivity, or intolerance to CB-012 or its excipients

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
(Part A) Number of patients with dose limiting toxicities (DLT) | 28 days
  Number of patients with DLTs during the 28 days following the first administration of CB-012.
(Part B) Overall Response Rate (ORR) | 12 months
  The ORR will be evaluated by European Leukemia Net (ELN) criteria

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - The University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - The Blood & Marrow Transplant Group of Georgia (BMTGA), Atlanta, Georgia
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - TriStar Bone Marrow Transplant, LLC, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin